CLINICAL TRIAL: NCT06722521
Title: Comparison of Intensive Lipid-Lowering Therapy With a Statin-Ezetimibe Combination (Without Aspirin) vs. Statin Monotherapy (With Aspirin) In Asymptomatic Patient With Coronary Artery Calcification
Brief Title: GUIDE-CAC: Statin-Ezetimibe Without Aspirin vs. Statin Monotherapy With Aspirin in High Coronary Calcification
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Seung-Whan Lee, M.D., Ph.D., Principal Investigator, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0193
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Primary Prevention; Vascular Calcification
Keywords: Cardiovascular Diseases; Aspirin; Statin
MeSH Terms: conditions — Vascular Calcification; Cardiovascular Diseases | interventions — pitavastatin; Ezetimibe; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive lipid-lowering therapy without aspirin (Experimental): In this group, intensive lipid-lowering therapy is performed without aspirin using pitavastatin 4 mg/ezetimibe 10 mg, targeting patients with coronary artery calcification (Agatston score ≥100) who require primary prevention and do not have physiologically significant coronary artery disease.
  ◦ Intervention Medications: Pitavastatin 4 mg/ezetimibe 10 mg (aspirin excluded)
  Interventions: Drug: Pitavastatin 4mg and ezetimibe 10mg, taken once daily
- Statin Monotherapy with Aspirin (Active Comparator): IIn this group, moderate-intensity lipid-lowering therapy is administered using pitavastatin 2 mg and aspirin for patients with coronary artery calcification (Agatston score ≥100) who require primary prevention and do not have physiologically significant coronary artery disease.
  ◦ Intervention Medications: Pitavastatin 2 mg and aspirin (Based on the clinician's judgment, the statin dosage may be increased to pitavastatin 4 mg depending on the LDL response, and if there are adverse effects associated with aspirin, it can be replaced with clopidogrel.)
  Interventions: Drug: Pitavastatin 2 mg with aspirin 100 mg, taken once daily.

INTERVENTIONS:
Drug: Pitavastatin 4mg and ezetimibe 10mg, taken once daily — Intensive lipid-lowering therapy without aspirin
  Arms: Intensive lipid-lowering therapy without aspirin
Drug: Pitavastatin 2 mg with aspirin 100 mg, taken once daily. — Moderate-intensity lipid-lowering therapy with aspirin
  Arms: Statin Monotherapy with Aspirin

SUMMARY:
A Multicenter, randomized trial comparing the efficacy and safety of intensive lipid-lowering therapy using a statin-ezetimibe combination without aspirin versus statin monotherapy with aspirin in asymptomatic patients with coronary artery calcification

DETAILED DESCRIPTION:
Coronary artery calcification is a well-established marker of subclinical atherosclerosis that effectively identifies high-risk individuals for cardiovascular events, even in asymptomatic patients. However, the optimal intensity of preventive interventions-particularly regarding the balance between efficacy and safety-remains unclear in asymptomatic patients with significant coronary calcification.

While aspirin has traditionally been used for the primary prevention of cardiovascular events, recent evidence suggests that its routine use in asymptomatic individuals may carry greater bleeding risks than cardiovascular benefits. In contrast, intensive lipid-lowering therapy with statins and ezetimibe has proven effective in reducing LDL-C levels and preventing cardiovascular events by slowing atherosclerotic progression and stabilizing plaques.

This study aims to evaluate whether intensive lipid-lowering therapy using a statin-ezetimibe combination (without aspirin) is non-inferior to statin monotherapy (with aspirin) in reducing cardiovascular events among patients with significant coronary artery calcification. By comparing these two strategies, we seek to establish whether more aggressive lipid management might obviate the need for aspirin in these intermediate- to high-risk yet asymptomatic patients.

ELIGIBILITY:
Inclusion Criteria

1. Adults aged 19 years and older
2. Asymptomatic patients with significant coronary calcification (Agatston score ≥ 100) and no physiologically significant coronary artery disease (CAD)

   * The coronary CT scan used to establish the CAC score must be performed within 3 years prior to randomization.
   * The assessment of physiological significance must be performed within 6 months prior to randomization
3. Participants will be eligible for inclusion regardless of prior statin or anti-platelet agents use.

Exclusion Criteria

1. Major ASCVD events (clinically documented ASCVD)

   If at least one of the following criteria is present via patient history, physical examination, or medical records at the time of screening, the patient is not eligible:
   * Acute coronary syndrome (MI or unstable angina)
   * Coronary revascularization (PCI, CABG) or other arterial revascularization
   * Ischemic stroke (Not TIA)
   * Symptomatic peripheral arterial disease (history of claudication with ABI <0.90, or previous revascularization or amputation
2. Patients with physiologically significant CAD

   * Moderate to severe CAD (diameter stenosis >50%) on CCTA with positive strest test (thallium, treadmil, stress echocardiography)
   * Moderate to severe CAD (diameter stenosis >50%) on CAG with positive fractional flow reserve (FFR) < 0.8
3. Patients with familial hypercholesterolemia.
4. Patients with low-density lipoproteins cholesterol (LDL-C) ≥ 190 mg/dL regardless taking a statin or not.
5. Continuation of PCSK9 inhibitor is required during the clinical trial
6. Patients with chronic kidney disease (<eGFR 30mL/min/1.73m2)
7. Advanced liver disease (Child-Pugh B or C)
8. Hepatic disease or biliary tract obstruction, or significant hepatic enzyme elevation (ALT or AST > 5 times upper limit of normal).
9. History of gastrointestinal bleeding, peptic ulcer, or intracranial hemorrhage within 6 months prior screening
10. Patients with a history of organ transplantation who are on immunosuppressive therapy
11. Concurrent use of other medications that may increase bleeding risk such NOAC and warfarin
12. A history of significant allergic reaction to aspirin or statin/ezetimibe
13. A diagnosis of cancer (other than superficial squamous or basal cell skin cancer) in the past 3 years or current treatment for the active cancer.
14. Life expectancy < 1 years for any non-cardiac or cardiac causes.
15. Patient's pregnant or breast-feeding or child-bearing potential.
16. Any clinically significant abnormality identified at the screening visit, physical examination, laboratory tests, or electrocardiogram which, in the judgment of the Investigator, would preclude safe completion of the study.
17. Unwillingness or inability to comply with the procedures described in this protocol

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7435 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2032-06-30 (Estimated); Study Completion 2032-10-31 (Estimated)

PRIMARY OUTCOMES:
Event rate of a major adverse cardiovascular events | 48months
  Death from any cause, myocardial infarction, stroke, urgent coronary revascularization, resuscitated cardiac arrest, or unstable angina related hospitalization

SECONDARY OUTCOMES:
Event rate of a all cause death | 48months
  All-cause mortality was used instead of cardiac mortality to avoid potentially difficult adjudication of causes of death, especially given the relatively low expected mortality rate. In addition, the cause of death will be adjudicated as being due to cardiovascular causes, non-cardiovascular causes, or undetermined causes.
Event rate of a cardiovascular death | 48months
  includes death resulting from an acute myocardial infarction (MI), sudden cardiac death, death due to heart failure (HF), death due to stroke, death due to cardiovascular (CV) procedures, death due to CV hemorrhage, and death due to other CV causes
Event rate of a spontaneous myocardial infarction | 48months
  A spontaneous myocardial infarction related to atherosclerotic plaque rupture, ulceration, fissuring, erosion, or dissection, resulting in intraluminal thrombus in one or more of the coronary arteries
Event rate of a stroke | 48months
  A. Ischemic Stroke B. Hemorrhagic Stroke C. Undetermined Stroke
Event rate of a urgent coronary revascularization | 48months
  1. Elective:
  2. Urgent:
  3. Emergency:
  4. Salvage:
Event rate of a Resuscitated cardiac arrest | 48months
Event rate of a unstable angina related hospitalization | 48months
Event rate of a composite of hard outcomes (all cause death, myocardial infarction and ischemic stroke) | 48months
Event rate of a Clinically relevant bleeding (Bleeding Academic Research Consortium definition ≥ type 2) | 48months
  Bleeding Academic Research Consortium definition ≥ type 2
Changes of Lipid profile | 48months
Treatment-emergent Serious Adverse Events resulting in Study Drug Discontinuation | 48months
  Liver function abnormalities(AST or ALT > 5x ULN)
  Renal function abnormalities (serum creatinine increase ≥3-fold from baseline OR increase to ≥4.0 mg/dL OR initiation of renal replacement therapy)
  Muscle-related events (Statin-associated muscle symptoms OR CK >5x ULN) (CK reference range: 50-250 IU/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea